CLINICAL TRIAL: NCT02687646
Title: Clinical Trial Phase I / II Graft Versus Host Disease Treatment Refractory to First-line Therapy With Sequential Infusion of Mesenchymal Cells Allogeneic Expanded Adipose Tissue in Vitro
Brief Title: Clinical Trial With MSC for Graft Versus Host Disease Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Andalusian Initiative for Advanced Therapies (Other Government)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC-EICH-2014; 2014-005533-32 (EudraCT Number)
Record Dates: First submitted 2016-01-19; First posted 2016-02-22 (Estimated); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Acute Graft Versus Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogeneic Mesenchymal Cells (Experimental): All patients will receive Adult Allogeneic Mesenchymal Cell from adipose tissue. It is not considered ethical the inclusion of a control group.
  Interventions: Drug: Adult Allogeneic Mesenchymal cells from adipose tissue.

INTERVENTIONS:
Drug: Adult Allogeneic Mesenchymal cells from adipose tissue. — Study treatment consists of Mesenchymal Stem Cell (MSC) derived from donors adipose tissue and expanded in vitro in a specific medium with platelet lysate without addition of animal derived products.
  Subjects will receive four sequential IV dose of Mesenchymal stem cells.
  Sequential doses:
  Day 1: 0.7-1 x 106 MSC / kg Day 4: 0.7-1 x 106 MSC / kg Day 11: 0.7-1 x 106 MSC / kg Day 18: 0.7-1 x 106 MSC / kg
  Other Names: MSC for the treatment of graft -versus -host disease

SUMMARY:
Sequential administration of MSCs obtained from adipose tissue is an effective and safe treatment for acute graft versus host disease refractory to first-line treatment. Furthermore the infusion of these cells produces a biological pattern in patients that relates to the clinical response.

DETAILED DESCRIPTION:
Multicenter, open, non -controlled clinical trial. It is a phase I-II trial to assess the safety and efficacy of sequential infusion of allogeneic MSCs from adipose tissue, expanded "in vitro" platelet lysate in the treatment of patients undergoing hematopoietic stem cell trasplantation, who have developed a refractory graft versus host disease to first line of treatment.

This is a prospective, multicenter, open to patients undergoing allogeneic transplantation in Spanish hospitals, with one cohort of patients who receive four sequential doses of MSC.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ≥ grade II Graft Versus Host Disease refractory to first-line treatment.
2. Having been subjected to hematopoietic Stem Cell Transplantation as treatment for malignant blood disorder has been controlled by the transplantation. The source may have been bone marrow cells or peripheral blood (PB) and coming from a family member or unrelated donor.
3. Having been transplanted with myeloablative or non-myeloablative conditioning.
4. normal cardiac function (EF ≥ 40%) without evidence of uncontrolled hypertension, congestive heart failure, angina pectoris or myocardial infarction within 6 months prior to the process
5. Lung function without evidence of severe obstructive or restrictive lung disease.
6. Age between 18 and 65 years.
7. Women of childbearing age considered until one year after the last menstrual period and which have not undergone a surgical sterilization must obtain a negative pregnancy test at the time of inclusion in the study and commit to use a medically approved birth control while on study.
8. normal cardiac function (EF ≥ 40%) without evidence of uncontrolled hypertension, congestive heart failure, angina pectoris or myocardial infarction within 6 months prior to the process.
9. Signature of informed consent -

Exclusion Criteria:

1. uncontrolled blood disorder by transplantation or progression at the time of inclusion.
2. bacterial, viral, fungal or is not being controlled.
3. Any circumstance that the proposed trial dissuade medical treatment. Pregnancy, lactation or refusal to use safe contraceptive measures.
4. Patients who are currently participating or have completed their participation in a clinical trial in less than 3 months or who have participated in a clinical trial of Advanced Therapies at any previous time period.
5. Patients who are currently participating or have completed their participation in a clinical trial in a period shorter than 3 months or who have participated in a clinical trial of Advanced Therapies at any previous time.
6. positive serology for Hepatitis B , Hepatitis C and AIDS Virus. -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Safety measured by incidence of serious adverse events | 2 years
  Safety will be measured in terms of:
  Incidence of Serious Adverse Events after at the time of the infusion of study drug or during follow-up.

SECONDARY OUTCOMES:
Effectiveness measured by answer of refractory acute graft disease against host to first-line treatment | 2 years
  Effectiveness will be measured in terms of:
  Answer of refractory acute graft disease against host to first-line treatment

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Caballero, Hematologist, Study Director — Virgen del Rocio University Hospital
Locations (6):
- Spain (6):
  - Clinica Universitaria de Navarra, Av Pio XII ,36, Pamplona, Navarre
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital clinico universitario de salamanca, Salamanca
  - Virgen del Rocio University Hospital, av. Manuel Siurot s/n, Seville

IPD SHARING:
Plan to Share IPD: Undecided